CLINICAL TRIAL: NCT02422238
Title: Disease Mechanisms and Markers for Non-alcoholic Steatohepatitis in a Population With Non-alcoholic Fatty Liver Disease: a Prospective Cohort Study With Biobank
Brief Title: Prospective Cohort, With Biobanking, of Patients With Nonalcoholic Fatty Liver Disease
Acronym: NAFLD-cohort
Status: Recruiting | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Centrum Obesitas-Eetstoornissen (CO-EUR) (Unknown)
Responsible Party: Principal Investigator, Ger Koek, MD, PhD, Maastricht University Medical Center
Other Study IDs: METC142074
Record Dates: First submitted 2015-04-16; First posted 2015-04-21 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Nonalcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine, faeces and exhaled air will be collected. The buffy coat of blood collected in an EDTA-tube to obtain plasma, will be stored for isolation of DNA.
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the present prospective NAFLD cohort study (with biobank), of obese subjects with proven NAFLD based on liver biopsy and/or MRI, is to study factors contributing to the development of NASH in patients with simple steatosis and to identify and validate non-invasive markers for the diagnosis of NASH.

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) is with 20-30% the most prevalent liver disorder in Western society. Most patients with NAFLD have no or few, mainly aspecific symptoms; and generally there is a silent progression of simple steatosis to NASH and in the end liver-related morbidity and mortality.

Further insight in factors contributing to the initiation of NASH in patients with simple steatosis and early diagnosis are essential for identifying future therapeutic options and to limit the risk of complicated NASH (i.e. fibrosis, and cirrhosis with portal hypertension) HCC, liver-related mortality and extrahepatic morbidity.

This cohort study, with both a cross-sectional and a longitudinal part, will include obese subjects (BMI ≥ 30 kg/m2, age 18-65) with proven NAFLD based on liver biopsy and/or MRI.

All participants will be asked to complete several questionnaires (i.e. demographics, clinical data, SF-36, GAD-7 and PHQ-9, FFQ, SQUASH, and Baecke), and to undergo anthropometric measurements. Furthermore, blood, urine, faeces and exhaled air will be collected and a fibroscan and DEXA-scan will be performed. Additionally, participants will be asked to participate in a multi-sugar test for intestinal permeability.

The majority of eligible subjects will undergo/have undergone a MRI or liver biopsy for clinical reasons. It is to be expected that about 33% of subjects will be asked to undergo a MRI for study purpose only.

After 5 and 10 years, participants will be invited to undergo in the same study procedures, data and sample collection to study the factors responsible for the development of NASH in the group with simple steatosis at baseline, and the development of (extra)hepatic complications in the group with NASH at baseline.

ELIGIBILITY:
Inclusion Criteria:

* NAFLD diagnosis based on evidence of hepatic steatosis, either by imaging (using MRI) or by histology.
* BMI ≥ 30 kg/m2
* Between 18 - 65 years of age

Exclusion Criteria:

* Incompetent to understand and/or sign the informed consent.
* Causes for secondary hepatic fat accumulation such as significant alcohol consumption, medications, Wilson's disease, viral infections, starvation or parenteral nutrition, among others, and conditions associated with microvesicular steatosis
* Ethanol consumption exceeding more than 14 standard beverages per week for males and more than 7 standard beverages per week for female.
* Not able or willing to undergo MRI (for example claustrophobia, ICD, pacemaker).
* Not willing to be informed about unexpected findings by MRI
* Unwilling to collect bio samples.
* Pregnancy and breastfeeding.
* Indication or planned for bariatric surgery within one year after inclusion or a history of bariatric surgery.
* Diagnosis of liver cirrhosis and/or hepatocellular carcinoma.
* Current diagnosis of extrahepatic malignancy(s) or prior diagnosis within last 5 years.
* Individuals about to undergo or recovering from a surgical or otherwise medical procedure that will interfere with data collection and analyses planned within the current cohort, will initially be excluded from participation, but are offered the opportunity to participate at a later moment in time

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese ( BMI ≥ 30 kg/m2) subjects with proven NAFLD either by imaging (using MRI) or histology, referred to secondary or tertiary care for obesity related problems will be asked to participate in this study.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Development of NASH | 10 years

SECONDARY OUTCOMES:
Prevalence of hepatic complications of NAFLD | 10 years
Prevalence of extrahepatic complications of NAFLD | 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Shami GJ, Samarska IV, Koek GH, Li A, Palma E, Chokshi S, Wisse E, Braet F. Giant mitochondria in human liver disease. Liver Int. 2023 Nov;43(11):2365-2378. doi: 10.1111/liv.15711. Epub 2023 Aug 24. PMID 37615254